CLINICAL TRIAL: NCT00890903
Title: Usage of Vinorelbin ORAL (Navelbine® ORAL) in the Treatment of Advanced Non-small Cell Lung Cancer(NSCLC)and Advanced Breast Cancer
Brief Title: Non-Interventional Study With Vinorelbine ORAL in Advanced Non-Small Cell Lung Carcinoma(NSCLC) and Metastatic Breast Cancer (MBC)
Status: Completed | Type: Observational
Sponsor: Pierre Fabre Pharma GmbH (Industry)
Collaborators: iOMEDICO AG (Industry)
Responsible Party: Sponsor
Other Study IDs: IOM-155
Record Dates: First submitted 2009-04-29; First posted 2009-04-30 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Non Small Cell Lung Carcinoma; Metastatic Breast Cancer
Keywords: NSCLC; non small cell lung carcinoma; metastatic breast cancer; MBC; advanced breast cancer; Navelbine; Navelbine-ORAL; Vinorelbine; Vinorelbine-ORAL; daily routine; concomitant antiemetic therapy; patient compliance; germany; non-interventional study; oral anti cancer therapy; quality of life
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Breast Neoplasms; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- NSCLC: Patients with advanced non-small cell lung cancer
- MBC: Female patients with metastatic, Anthracycline-resistent breast cancer

SUMMARY:
The purpose of this non-interventional study is to collect data on efficacy and toxicity of the use of Navelbine ORAL in daily routine in Germany (especially after availability of an 80mg capsule). The study focusses on concomitant antiemetic therapy and patient compliance.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Male and female patients
* Advanced NSCLC (Stage III or IV) or Antracycline-resistant MBC
* Therapy with Navelbine capsules in any palliative treatment line
* Signed patient informed consent

Exclusion Criteria:

* Pregnancy and nursing
* All other exclusion criteria listed in SPC (summary of product characteristics)
* lack of signed Patient informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced non-small cell lung cancer (NSCLC) or metastatic, Antracycline-resistant breast cancer, treated with Navelbine capsules
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2009-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Progression-free-survival | 1 year after LPI

SECONDARY OUTCOMES:
Time to progression | 1 year after LPI
Adverse reactions | 1 year after LPI
Concomitant antiemetic therapy | 1 year after LPI
Patient compliance | 1 year after LPI
Recording of combinations of applied capsules (requested by a patients' questionnaire) | 1 year after LPI
General condition of patients (requested by a patients' questionnaire) | 1 year after LPI
Therapy performance in the daily routine | 1 year after LPI

CONTACTS AND LOCATIONS:
Locations (1):
- Pierre Fabre Pharma GmbH, Freiburg im Breisgau, Germany